CLINICAL TRIAL: NCT04724668
Title: The Role of the Circadian System in Binge Eating Disorder
Acronym: CHRONO-BE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Lindner Center of HOPE (Other)
Responsible Party: Principal Investigator, Francisco Romo-Nava, Associate Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2020-0345; 1K23MH120503-01A1 (NIH)
Record Dates: First submitted 2021-01-20; First posted 2021-01-26 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Binge-Eating Disorder; Circadian Rhythm Disorders
Keywords: Binge eating; Circadian
MeSH Terms: conditions — Binge-Eating Disorder; Chronobiology Disorders; Bulimia | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: The specific aims will be completed in a two-phase experimental approach. In the first phase (specific aim 1), subjects with obesity with BED (n=40) and without BED (n=40) will participate in a 2-week longitudinal study. In the second phase (specific aim 2), only BED subjects that complete phase 1 will rollover for a 4-week intervention study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: On the intervention phase 2 (Specific aim 2). Only subjects with BED (n=40) will participate and be randomly assigned to one of two combinations of morning lights and/or melatonin/placebo (20 subjects/each arm). Researchers and participants will be blinded to the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Morning light version+ Melatonin (Other): Morning light version and melatonin 3mg capsule (3hrs before DLMO)
  Interventions: Dietary Supplement: Melatonin (3hrs before DLMO); Device: Morning light version 1
- Morning light version+ Placebo (Other): Morning light version and placebo capsule (3hrs before DLMO)
  Interventions: Dietary Supplement: Placebo (3hrs before DLMO); Device: Morning light version 2

INTERVENTIONS:
Dietary Supplement: Melatonin (3hrs before DLMO) — Melatonin 3mg (3hrs before DLMO)
  Arms: Morning light version+ Melatonin
Dietary Supplement: Placebo (3hrs before DLMO) — Placebo capsule (3hrs before DLMO)
  Arms: Morning light version+ Placebo
Device: Morning light version 1 — Morning light version
  Arms: Morning light version+ Melatonin
Device: Morning light version 2 — Morning light version
  Arms: Morning light version+ Placebo

SUMMARY:
Binge eating disorder (BED) shows prominent circadian features that suggest a delay in circadian phase, and preliminary evidence shows binge eating may be responsive to chronobiological interventions, implicating a circadian system dysfunction in its pathophysiology. What remains lacking, however, is comprehensive knowledge of the characteristics of circadian system dysfunction in BED, and whether this dysfunction represents a therapeutic target in BED. There is therefore a critical need to characterize circadian system dysfunction in BED, and evaluate it as a potential therapeutic target. Without such information, the understanding on the role of the circadian system in BED and its potential as a new therapeutic target will remain limited.

DETAILED DESCRIPTION:
The overall objective of the research strategy will be to characterize circadian system dysfunction in BED and its potential as a therapeutic target. The central hypothesis is that a circadian system dysfunction (phase delay) plays a role in the pathophysiology of BED, and that advancing the circadian phase will improve BED symptoms. To attain the overall objectives, the following specific aims will be pursued in two phases:

Specific aim 1) To characterize circadian system dysfunction in BED (Phase 1). Circadian system function will be evaluated in 80 adult (18 to 50yrs) obese subjects, 40 with BED and 40 without BED as a control group matched by age, body mass index (BMI), and gender, during a two-week observational phase. Based on preliminary data, the working hypothesis is that DLMO (the primary outcome measure) and secondary circadian parameters (i.e., locomotor activity acrophase) will occur later in the BED group compared with the control group, and a later circadian phase will be associated with worse BED clinical features.

Specific aim 2) To evaluate circadian phase as a predictive biomarker for response to a chronobiological intervention and evidence of circadian system target engagement in BED (Phase 2). A mechanistic clinical trial with a 4-week double-blinded, randomized, sham/placebo controlled study design will evaluate the effect of a combination of morning lights+Melatonin/placebo on the circadian system and eating behavior on 40 BED subjects that complete phase 1. Subjects will be randomized to receive a combination of morning lights at usual wake time + Melatonin(3mg) or placebo (3hr before DLMO). Based on preliminary data, the working hypothesis is that a chronobiological intervention will induce a greater DLMO advance (primary outcome measure), greater decrease in binge eating days/week (secondary outcome measure), and change in exploratory metabolic outcomes. In addition, a later baseline DLMO (secondary outcome) will predict change in binge eating days/week and metabolic parameters in response to a chronobiological intervention.

ELIGIBILITY:
Binge Eating Disorder (BED) group inclusion criteria:

1. Age 18-50 years, inclusive
2. Female or male
3. BMI ≥30 kg/m2
4. Current BED diagnoses by Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) criteria confirmed by Structured Clinical Interview (SCID-5)
5. Moderate or severe BED (≥3 binge eating episodes/week in the past 14 days)
6. No current pharmacological treatment for BED, or if receiving treatment dose stable for ≥ 2 months
7. If receiving psychotherapy, intervention must be stable for ≥ 3 months and agree to continue during the study
8. Other psychiatric disorders will be permitted as long as they are not more than moderate in severity
9. Using an effective contraceptive method (participants of childbearing potential)

BED exclusion criteria:

1. Current severe comorbid psychopathology (i.e; mania, severe major depressive disorder (MDD), psychosis)
2. Current (past month) substance use disorder (caffeine and nicotine allowed)
3. Chronic use of bright light therapy (BLT) or melatonin in the past month
4. Current contraindication or history of melatonin allergy or non-tolerability;
5. Current contraindication or history of BLT non-tolerability
6. Significant risk of suicide according to Columbia-Suicide Severity Rating Scale (CSSRS) or clinical judgment, or suicidal behavior in the past year
7. Routine shift work (night work) in the past month
8. Travel across more than 1 time zone in the past two weeks
9. Current treatment with medication known to affect the circadian system or melatonin measurements, including: B-blockers, hypnotic sedatives, anticoagulants, antidiabetes drugs, oral corticosteroids, and other immunosuppressant medication
10. Current lesions or bleeding in the oral cavity, as it may alter DLMO measurements
11. Clinically significant unstable medical conditions as judged by the clinician, including: seizure or neurodegenerative disorders, thyroid conditions, autoimmune disorders, and cardiovascular disease
12. Pregnancy or breastfeeding
13. Participation in a clinical trial in the past month
14. Suspected intelligence quotient (IQ) <80
15. Any other clinically relevant reason as judged by the clinician

Control group inclusion criteria:

1. Age 18-50 years, inclusive
2. Female or male;
3. BMI ≥30 kg/m2
4. No current or lifetime history of BED or bulimia nervosa diagnoses confirmed by SCID-5
5. No current (past month) psychiatric diagnosis according to SCID-5, including substance use disorders (caffeine and nicotine allowed)
6. No current psychiatric or psychological treatment, or if receiving treatment dose/intervention stable for ≥ 2 months

Control group exclusion criteria:

1. Clinically significant unstable medical conditions as judged by the clinician, including: seizure or neurodegenerative disorders, thyroid conditions, autoimmune disorders, and cardiovascular disease
2. Chronic treatment with BLT or melatonin in the past month
3. Routine shift work (work at night) in the past month
4. Travel across more than 1 time zone in the past two weeks
5. Significant risk of suicide according to CSSRS or clinical judgment, or suicidal behavior in the past year
6. Current treatment with medication known to affect the circadian system or melatonin measurements, including, B-blockers, hypnotic sedatives, anticoagulants, antidiabetes drugs, oral corticosteroids, and other immunosuppressant medication
7. Current lesions or bleeding in the oral cavity, as it may alter DLMO measurements
8. Pregnant or breastfeeding
9. Participation in a clinical trial in the past month
10. Suspected IQ<80
11. Any other clinically relevant reason as judged by the clinician

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Phase 1 Dim Light Melatonin Onset (DLMO) | Phase 1 baseline (visit 0)
  Difference in mean DLMO (measured in time) between subjects with binge eating disorder (BED) and control subjects without BED.
Phase 2 Dim Light Melatonin Onset (DLMO) | Phase 2 baseline (visit 0) to endpoint, on average one month.
  Differences in DLMO (measured in time) change from baseline to endpoint between two intervention groups will be analyzed using an ANCOVA model with age as a covariate.

SECONDARY OUTCOMES:
Phase 1 Locomotor activity acrophase | Phase 1 baseline (visit 0)
  Difference in mean locomotor activity acrophase (7 days) measured in time between BED and control subjects without BED
Phase 1 Midline Estimating Statistic of Rhythm (MESOR) | Phase 1 baseline (visit 0)
  Difference in mean MESOR (7 days) measured in time between BED and control subjects without BED
Phase 1 MEQ | Phase 1 baseline (visit 0)
  Difference in mean Morningness Eveningness Questionnaire scores (MEQ) between BED and control subjects without BED. MEQ score range 18 to 86, lower scores indicate more eveningness, higher scores indicate more morningness.
Phase 1 Association between DLMO and binge eating days/week | Phase 1 baseline (visit 0)
  The association between DLMO (measured in time) and binge eating days/week in BED subjects.
Phase 2 Binge eating days/week | Phase 2 baseline (visit 0) to endpoint, on average one month.
  Differences in Binge eating days/week from baseline to endpoint between groups will be analyzed using an ANCOVA model with age as a covariate.
Phase 2 Locomotor activity acrophase | Phase 2 baseline (visit 0) to endpoint, on average one month.
  Differences in locomotor activity acrophase from baseline to endpoint between groups will be analyzed using an ANCOVA model with age as a covariate.
Phase 2 baseline (visit 0) to endpoint | Phase 2 baseline (visit 0) to endpoint, on average one month.
  Differences in MESOR (Midline Estimating Statistic of Rhythm) from baseline to endpoint between groups will be analyzed using an ANCOVA model with age as a covariate.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Romo-Nava, MD, PhD, Principal Investigator — University of Cincinnati/ Lindner Center of HOPE
Locations (1):
- Lindner Center of HOPE / University of Cincinnati, Mason, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
However, individual participant data may be shared with other researchers upon request.